CLINICAL TRIAL: NCT00143351
Title: Open Extension Study Evaluating the Long-term Efficacy, Safety, and Tolerability of Oral Ziprasidone in the Treatment of Resistant/Intolerant Schizophrenic Patients Who Have Acutely Responded to Ziprasidone in the Mozart Study
Brief Title: Mozart Relapse Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281088
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone

INTERVENTIONS:
Drug: Ziprasidone

SUMMARY:
To assess the long-term efficacy of oral Ziprasidone in the maintenance treatment of resistant schizophrenic subjects who have benefited from participation in the phase III ziprasidone study A1281039 (MOZART study), to assess the efficacy of ziprasidone in the relapse prevention of schizophrenia, to collect long-term data on safety and tolerability of oral Ziprasidone

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed MOZART study and who are responders to Ziprasidone:
* Responders: patients with a 20% or more reduction in the PANSS total score at the endpoint of the Mozart Study (recorded at V18 in the Mozart) as compared with the baseline value
* Patients not hospitalised in an acute psychiatric service
* Written, informed consent to participation.
* Female patients of at risk of pregnancy must avoid to remain pregnant; if already used, an adequate method of contraception can be continued

Exclusion Criteria:

* Psychiatric:
* Subjects with a score of greater than or equal to 5 and an increase of at least 2 points (with respect to baseline value of MOZART study) at one of the following PANSS items: P7 (hostility), G8 (uncooperativeness) or G14 (poor control impulse)
* Subjects with a score equal to 3 and an increase of at least 1 point (with respect to baseline value of MOZART study) at item 8 (suicide) of CDSS
* General:
* Patients who, during MOZART study, have developed one of the following diseases will be excluded: (or patients who do not satisfy anymore one of the following general exclusion criteria of MOZART study)
* Subjects with a history of clinically significant and/or currently relevant haematological, renal (including single kidney), hepatic, gastrointestinal, endocrine (except for current adequately treated hypo- or hyperthyroidism), pulmonary (excluding chronic bronchitis, mild emphysema or chronic obstructive pulmonary disease), dermatological, oncological, or neurological disease, excluding tardive dyskinesia but including all forms of epilepsy (febrile convulsions in childhood acceptable). The only subjects with known prior malignant disease who are eligible are those with cured prior skin cancer. Controlled Type II diabetes (glucose < 180 mg/100 ml at screening and baseline with dietary or oral hypoglycemic treatment) will not be considered a significant medical illness and would not exclude a subject from the study
* Patients with a non stabilized somatic disease - Acute or chronic heart disease
* Clinically significant ECG abnormalities
* Subjects with QTc greater than or equal to 500 msec (subjects with QTc greater than or equal to 450 msec and < 500 msec should be discussed with the cardiologist) - Concomitant treatment with medications that prolong QTc interval (please review prescribing information of other treatments)
* Subjects with serum K+ outside the normal range
* History of seizure (should be discussed with the Sponsor)
* Subject with any confirmed laboratory values that deviate from the upper or lower limits of normal prior to study entry, except for clinically insignificant deviations as determined by investigator
* Pregnant or lactating women
* Subjects who intend to donate blood or blood products during the 4 weeks prior to the study, during the study or in the 30 days after the study ends
* Subjects unable or unlikely to follow the study protocol
* Subjects with a history of neuroleptic malignant syndrome developing from the administration of antipsychotic compounds
* Diagnosis of substance dependence using DSM-IV criteria (305.xx)
* Positive urine drug screen at screening for amphetamines, cocaine or opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2003-06; Study Completion 2005-09

PRIMARY OUTCOMES:
long-term efficacy of oral Ziprasidone in the maintenance treatment

SECONDARY OUTCOMES:
To assess the efficacy of ziprasidone in the relapse prevention of schizophrenia To collect long-term data on safety and tolerability of oral Ziprasidone

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Italy (14):
  - Pfizer Investigational Site, Vicenza, Bassano DEL Grappa
  - Pfizer Investigational Site, Città di Castello, Perugia
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Brescia
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Guardiagrele (CH)
  - Pfizer Investigational Site, Messina
  - Pfizer Investigational Site, Parma
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Sassari
  - Pfizer Investigational Site, Terni
  - Pfizer Investigational Site, Torino
  - Pfizer Investigational Site, Trieste
  - Pfizer Investigational Site, Verona